CLINICAL TRIAL: NCT01078337
Title: T-cell MRD Evaluation Using Flow Cytometric Analysis
Brief Title: T-cell Minimal Residual Disease (MRD) Evaluation Using Flow Cytometric Analysis
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Gary V Dahl, Stanford University School of Medicine
Other Study IDs: SU-11022007-790; PEDSALL0001
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia, Lymphocytic, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and bone marrow

INTERVENTIONS:
Procedure: bone marrow aspiration
Procedure: peripheral blood sampling

SUMMARY:
To determine if MRD (minimal residual disease) can be found in the blood (only) as opposed to bone marrow in children with ALL (acute lymphoblastic leukemia).

ELIGIBILITY:
Inclusion Criteria:

* Children with newly diagnosed T-cell ALL

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with newly diagnosed T-cell ALL
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2002-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary V Dahl, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States